CLINICAL TRIAL: NCT05302323
Title: Evaluation of the Effect of Surgical Drapes on Intraoperative Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neslihan Ilkaz (Other)
Responsible Party: Sponsor-Investigator, Neslihan Ilkaz, Operating Room Nurse, PhD, RN, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Organization: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Interventional
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Hypothermia
Keywords: Hypothermia; perioperative nursing; operating room nursing; unintended hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: major abdominal surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disposable Drapes (Other): group using disposable surgical drapes
  Interventions: Other: Disposable Drape
- Reusable Drapes (Other): group using reusable surgical drapes
  Interventions: Other: Reusable Drape

INTERVENTIONS:
Other: Disposable Drape — Disposable surgical drapes, consisting of 6 pieces, were used as a set during surgery
  Arms: Disposable Drapes
Other: Reusable Drape — Reusable surgical drapes, consisting of 6 pieces, were used as a set during surgery
  Arms: Reusable Drapes

SUMMARY:
This study was planned to investigate whether the wetness of surgical drapes (disposable and resusable drapes) used in the intraoperative period causes hypothermia.

DETAILED DESCRIPTION:
After being informed about the study and potential risk all patients giving written informed consent then the study started. Patients who will undergo elective, gastrointestinal and other major abdominal surgery were included in the study. After patients were randomized by the investigator, patients were covered with disposable or reusable surgical drapes in accordance with hospital procedure. The body temperatures of the patients were followed for 2-6 hours as tympanic and esophageal. In addition, pre- and postoperative surgical drapes, sponges, compresses were measured with precision scales.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2-3
* Patients with abdominal surgery
* Patients receiving general anesthesia

Exclusion Criteria:

* Unwanted to participate in the study
* Patients over 70 years of age
* Presence of central (high) fever originating from the central nervous system resulting from conditions such as cerebrovascular disease, cerebral trauma, intracranial surgery, epilepsy or acute hydrocephalus
* Abnormalities of thermoregulation such as hypothyroidism, hyperthyroidism, history of malignant hyperthermia, or neuroleptic malignant syndrome
* Presence of infectious fever
* ASA 4 and above
* Emergency surgery
* Patients receiving pre-operative chemotherapy
* Having problems such as tearing and perforation of the covers during the work.
* Patients being hyperthermic in the intraoperative process

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
tympanic and esophageal body temperature measurement between two groups | throughout the operation (min.2 hours) (max. 6 hours)
  Tympanic and esophageal body temperature measurement between the two groups was followed throughout the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane training and research hospital, Ankara, Keçiören, Turkey (Türkiye)

REFERENCES:
- [Background] Hooper VD, Chard R, Clifford T, Fetzer S, Fossum S, Godden B, Martinez EA, Noble KA, O'Brien D, Odom-Forren J, Peterson C, Ross J. ASPAN's evidence-based clinical practice guideline for the promotion of perioperative normothermia. J Perianesth Nurs. 2009 Oct;24(5):271-87. doi: 10.1016/j.jopan.2009.09.001. No abstract available. PMID 19853810
- [Background] Hooper VD, Chard R, Clifford T, Fetzer S, Fossum S, Godden B, Martinez EA, Noble KA, O'Brien D, Odom-Forren J, Peterson C, Ross J, Wilson L; ASPAN. ASPAN's evidence-based clinical practice guideline for the promotion of perioperative normothermia: second edition. J Perianesth Nurs. 2010 Dec;25(6):346-65. doi: 10.1016/j.jopan.2010.10.006. No abstract available. PMID 21126665
- [Background] Bashaw MA. Guideline Implementation: Preventing Hypothermia. AORN J. 2016 Mar;103(3):305-10; quiz 311-3. doi: 10.1016/j.aorn.2016.01.009. PMID 26924369
- [Background] NICE. Hypothermia: prevention and management in adults having surgery. Clinical guideline Published: 23 April 2008, Last Updated 2016, nice.org.uk/guidance/cg65
- [Background] Association of periOperative Registered Nurses. Recommended practices for selection and use of surgical gowns and drapes. AORN J. 2003 Jan;77(1):206-10, 213. doi: 10.1016/s0001-2092(06)61392-6. No abstract available. PMID 12575635
- [Background] Maglinger PE, Sessler DI, Lenhardt R. Cutaneous heat loss with three surgical drapes, one impervious to moisture. Anesth Analg. 2005 Mar;100(3):738-742. doi: 10.1213/01.ANE.0000143954.98285.63. PMID 15728062
- [Background] NICE. Inadvertent perioperative hypothermia Overview. http://pathways.nice.org.uk/pathways/inadvertent-perioperative-hypothermia. 27.11.2017
- [Background] Guideline Quick View: Hypothermia. AORN J. 2019 Oct;110(4):463-465. doi: 10.1002/aorn.12843. No abstract available. PMID 31560431